CLINICAL TRIAL: NCT00234858
Title: A Phase IV, Randomized, Open-Label, Active Controlled Study to Compare the Effects of Tarka® and Hyzaar® on Glucose Tolerance in Subjects With Metabolic Syndrome
Brief Title: Tarka vs. Hyzaar in Patients With Metabolic Syndrome (STAR)
Acronym: STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, MD, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M03-598
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension; Metabolic Syndrome
Keywords: Hypertension; Metabolic Syndrome; Tarka; Hyzaar
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — trandolapril; Verapamil; hydrochlorothiazide, losartan drug combination; Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: trandolapril/verapamil
- 2 (Active Comparator)
  Interventions: Drug: (Hyzaar) losartan/hydrochlorothiazide

INTERVENTIONS:
Drug: trandolapril/verapamil — 2/180 mg QD with titration if needed at Week 4 to 4/240 mg QD
  Other Names: ABT-TARKA; Tarka
  Arms: 1
Drug: (Hyzaar) losartan/hydrochlorothiazide — 50/12.5 mg QD with titration if needed at Week 4 to 100/25 mg QD
  Other Names: Hyzaar; losartan/hydrochlorothiazide
  Arms: 2

SUMMARY:
The primary objective of this study is to determine whether impaired glucose tolerance is improved to a greater degree by Tarka than Hyzaar in subjects with metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome
* Fasting blood glucose between 100 mg/dL and 125 mg/dL
* Hypertension
* One additional criteria, Exclusion 1

Exclusion Criteria:

* Subject has a current diagnosis of Type 1 or Type 2 diabetes mellitus.
* Subject has a hypersensitivity to ACE inhibitor, ARB, CCB, clonidine, methyldopa, hydralazine, or thiazide diuretic medication.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2004-03; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Oral Glucose Tolerance | up to 1 year / 52 weeks

SECONDARY OUTCOMES:
Changes in blood pressure (BP), pulse rate and BP control. HbA1c, insulin sensitivity, insulin release, albuminuria, lipid profile, AMBP, clinical safety labs and adverse events. | up to 1 year / 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott

REFERENCES:
- [Derived] Bakris G, Molitch M, Hewkin A, Kipnes M, Sarafidis P, Fakouhi K, Bacher P, Sowers J; STAR Investigators. Differences in glucose tolerance between fixed-dose antihypertensive drug combinations in people with metabolic syndrome. Diabetes Care. 2006 Dec;29(12):2592-7. doi: 10.2337/dc06-1373. PMID 17130190